CLINICAL TRIAL: NCT01445067
Title: Phase I, Open-Label, Randomized, Single Sequence Study With Two Dose Groups to Compare the Pharmacokinetics of BMS-927711 in Migraine Subjects During an Acute Migraine Attack and During Non-Migraine Period
Brief Title: Study to Evaluate the PK of BMS-927711 in Patient With Migraine During Acute Migraine and Non-migraine Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN170-004
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2022-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: BMS-927711 (300 mg) (Active Comparator)
  Interventions: Drug: BMS-927711 (CGRP Antagonist)
- Arm 2: BMS-927711 (600 mg) (Active Comparator)
  Interventions: Drug: BMS-927711 (CGRP Antagonist)

INTERVENTIONS:
Drug: BMS-927711 (CGRP Antagonist) — Capsule, Oral, 300 mg, Once, One day
  Arms: Arm 1: BMS-927711 (300 mg)
Drug: BMS-927711 (CGRP Antagonist) — Capsule, Oral, 600 mg, Once, One day
  Arms: Arm 2: BMS-927711 (600 mg)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of BMS-927711 during migraine and non-migraine condition.

DETAILED DESCRIPTION:
Study Classification: Safety CGRP = Calcitonin gene related peptide

ELIGIBILITY:
Inclusion Criteria:

* Patients with migraine with or without aura who are otherwise healthy as determined by medical history, physical examination, clinical laboratory evaluations and 12-lead electrocardiogram (ECG), will be eligible
* Men or women [women of childbearing potential (WOCBP) or Women of non childbearing potential (WONCBP)] ages 18-55 years inclusive, with a body mass index (BMI) of 18.0 to 32.0 kg/m2 with not more than 8 migraines a month
* Patient has at least 1 year history of migraines (with or without aura) including the following:

  1. Meet the diagnostic criteria for migraine with history of at least 1 year (with or without aura) at the screening visit
  2. Migraine attacks with the age of onset prior to 55 years old
  3. Migraine attacks, on average, lasts about 4-72 hours if untreated in the 3 months prior to screening visit
* 2-8 moderate or severe migraine attacks per month in the 3 months prior to screening visit. The migraine, for which the patient receives treatment during the study, must have at least one of the associated symptoms: nausea, photophobia, phonophobia, or migraine with aura

Exclusion Criteria:

* Female patient is pregnant/breast-feeding (or is a female expecting to conceive during study period)
* Patient has history or evidence of stroke/transient ischemic attacks, heart disease, coronary artery vasospasm, other significant underlying cardiovascular diseases, uncontrolled hypertension (high blood pressure), uncontrolled diabetes, or Human Immunodeficiency Virus (HIV)
* Patient will be excluded if they take medications for acute migraine more than 10 days per month, had very frequent chronic tension type headaches for 15 or more days per month (or were unable to distinguish between tension-type headaches and migraine)
* Patient has major depression, other pain syndromes that might interfere with study assessments, psychiatric conditions, dementia, or significant neurological disorders (other than migraine)
* Patient has a history of gastric, or small intestinal surgery, or has a disease that causes mal absorption
* Patient has a history or current evidence of any unstable medical conditions (eg, history of congenital heart disease or arrhythmia, known suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial
* Patient has basilar migraine and hemiplegic migraine
* Patient taking narcotic medication
* History of alcohol, substance or drug abuse within the last year
* Uses an opiate as first line acute treatment for migraine attacks
* History of ergotamine, any acute therapy or triptan intake on greater than/equal 10 days per month on a regular basis for greater than/equal 3 months
* History of simple analgesic intake on greater than/equal 10 days per month for greater than/equal 3 months
* History of use of opioid or combination medication intake or butalbital containing analgesic greater than 5 days per month for greater than/equal to 3 months
* Do not receive migraine relief from a triptan migraine treatment
* Evidence of renal impairment - calculated creatinine clearance <60ml/min or clinically relevant finding on urinalysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-927711 will be derived from plasma concentration versus time | PK samples will be collected for up to 24 hours after the dosing
Time of maximum observed plasma concentration (Tmax) of BMS-927711 will be derived from plasma concentration versus time | PK samples will be collected for up to 24 hours after the dosing
Area under the plasma concentration-time curve from time zero to 24 hours post dose [AUC(0-24)] of BMS-927711 will be derived from plasma concentration versus time | PK samples will be collected for up to 24 hours after the dosing
Observed plasma concentration at 0.5 hr (C0.5h) of BMS-927711 will be derived from plasma concentration versus time | PK samples will be collected for up to 24 hours after the dosing
Observed plasma concentration at 2h (C2h) of BMS-927711 will be derived from plasma concentration versus time | PK samples will be collected for up to 24 hours after the dosing
Apparent total body clearance (CLT/F) of BMS-927711 will be derived from plasma concentration versus time | PK samples will be collected for up to 24 hours after the dosing

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) will be derived from plasma concentration versus time | From Day 1 0 hour to Day 2 24 hour time points
  Individual subject pharmacokinetic parameter values will be derived by non compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses
Time of maximum observed plasma concentration (Tmax) will be derived from plasma concentration versus time | From Day 1 0 hour to Day 2 24 hour time points
  Individual subject pharmacokinetic parameter values will be derived by non compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses
Area under the plasma concentration-time curve from time zero to 24 hours post dose [AUC (0-24)] will be derived from plasma concentration versus time | From Day 1 0 hour to Day 2 24 hour time points
  Individual subject pharmacokinetic parameter values will be derived by non compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses
Observed plasma concentration at 0.5 hr (C0.5h) will be derived from plasma concentration versus time | From Day 1 0 hour to Day 2 24 hour time points
  Individual subject pharmacokinetic parameter values will be derived by non compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses
Observed plasma concentration at 2 hr (C2h) will be derived from plasma concentration versus time | From Day 1 0 hour to Day 2 24 hour time points
  Individual subject pharmacokinetic parameter values will be derived by non compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses
Apparent total body clearance (CLT/F) will be derived from plasma concentration versus time | From Day 1 0 hour to Day 2 24 hour time points
  Individual subject pharmacokinetic parameter values will be derived by non compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - California Clinical Trials Medical Group, Glendale, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Compass Research, Llc, Orlando, Florida
  - Community Research, Cincinnati, Ohio

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx